CLINICAL TRIAL: NCT00301080
Title: A Phase III Study of D-Cycloserine in the Management of Paclitaxel-Induced Peripheral Neuropathic Pain in Breast Cancer Patients
Brief Title: D-cycloserine in the Management of Chemotherapy-Induced Peripheral Neuropathic Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding for the study fell through.
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NU 05CC2; 504-038 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Neurotoxicity; Pain; Breast Cancer
Keywords: pain; neurotoxicity; breast cancer
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain; Breast Neoplasms | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (original version) (Placebo Comparator): Placebo administered orally twice per day for 4 weeks.
  Interventions: Other: Placebo
- D-cycloserine 200mg (Active Comparator): D-cycloserine administered orally at a dose of 200 mg twice per day for 12 weeks.
  Interventions: Drug: D-cycloserine
- D-cycloserine 50 mg (Active Comparator): D-cycloserine administered orally at a dose of 50 mg twice per day for 12 weeks.
  Interventions: Drug: D-cycloserine
- D-cycloserine 250mg (Active Comparator): This was the original active comparator arm (before the design was changed): D-cycloserine administered orally at a dose of 250 mg twice per day for 4 weeks.
  Interventions: Drug: D-cycloserine
- Placebo (revised version) (Placebo Comparator): Placebo administered orally twice per day for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: D-cycloserine
  Other Names: Cycloserine; Seromycin™
  Arms: D-cycloserine 200mg; D-cycloserine 250mg; D-cycloserine 50 mg
Other: Placebo
  Arms: Placebo (original version); Placebo (revised version)

SUMMARY:
D-cycloserine may help lessen pain and other symptoms of peripheral neuropathy caused by chemotherapy. It is not yet known whether D-cycloserine is more effective than a placebo in treating peripheral neuropathy caused by chemotherapy.

This randomized, double-blind, placebo-controlled clinical trial was designed to study D-cycloserine at 2 different doses to see how well each works compared to the other and to a placebo in treating cancer patients with peripheral neuropathy caused by chemotherapy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study. Initially, patients were randomized to 1 of 2 treatment arms (D-cycloserine 250 mg twice daily or placebo twice daily), and treated for up to 4 weeks in the absence of unacceptable toxicity.

Later, the design was changed to randomize patients to 1 of 3 arms as follows:

* D-cycloserine 50 mg twice daily for up to 12 weeks
* D-cycloserine 200 mg twice daily for up to 12 weeks
* Placebo twice daily for up to 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients will be at least 18 years of age.
* Patients will be experiencing moderate to severe peripheral neuropathic pain
* Patients may be on chronic adjuvant pain medications such as antidepressants but must be on stable doses for at least one week prior to admission.
* Patients may be taking concurrent opioids but they must be willing to allow us to monitor their opioid use while on the trial.
* Patients must have chronic peripheral neuropathic pain will be defined as pain of 3 or more months duration which began in association with chemotherapy.
* Patient's will have bilateral peripheral neuropathic pain symptoms primarily involving the feet
* Patients must have breast cancer (any stage)
* Patients must be able to read and speak English and provide informed consent.
* Patients may be receiving chemotherapy as long as the agents are not known to cause a peripheral neuropathy.
* Patients must have an ECOG Performance Status < 3 and be able to attend the physician study visits
* Patients must not concurrently use gabapentin or pregabalin or must be willing to wean off their anti-convulsant medications prior to starting the trial.
* Patients may have diabetes mellitus (type 1 or 2) as long as there is no preexisting neuropathy.

Exclusion criteria:

* Patients will not have secondary cause of neuropathic pain including: HIV/AIDS,traumatic injury, or a personal history of non chemotherapy-induced neuropathy.
* Patients will not have a history of major depression or severe anxiety.
* Women of childbearing age will agree to take measures to prevent pregnancy and will not breast-feed while on the study medication. Women who are currently pregnant will not be invited to participate in this study.
* Patients will not have a history of seizures.
* Patients cannot be currently receiving antibiotic therapy for tuberculosis (e.g. isoniazid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Paice, PhD, RN, Principal Investigator — Northwestern University; Jamie Von Roenn, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Wisconsin School of Medicine, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened in 02/2006 (2-arm design with a 4 week treatment period). The 1st patient enrolled in 05/2006; 7 patients enrolled before it was suspended in 04/2007 pending revision (new 3-arm design & 12 week treatment period). Re-opened in 09/2007, but drug manufacturing & funding issues forced it to terminate with no further accrual in 05/2008.
Groups:
- Placebo (Original Version): Placebo administered orally at a dose of twice per day for 4 weeks.
- Placebo (Revised Version): Placebo administered orally at a dose of twice per day for 12 weeks.
Period: Original Version (2 Arms & 4 Weeks)
Arm/Group | D-cycloserine 250mg | Placebo (Original Version) | D-cycloserine 200mg | D-cycloserine 50 mg | Placebo (Revised Version)
Started | 4 | 3 | 0 (This arm not part of the original version.) | 0 (This arm not part of the original version.) | 0 (This arm not part of the original version.)
Received an Intervention | 3 | 3 | 0 | 0 | 0
Completed 4 Week Intervention | 3 | 3 | 0 | 0 | 0
Completed | 3 | 3 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Never received drug | 1 | 0 | 0 | 0 | 0
Period: Revised Version (3 Arms & 12 Weeks)
Arm/Group | D-cycloserine 250mg | Placebo (Original Version) | D-cycloserine 200mg | D-cycloserine 50 mg | Placebo (Revised Version)
Started | 0 (This arm was not a part of the revised study design.) | 0 (This arm was not a part of the revised study design.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants (Original Version): All 7 patients enrolled were during the original version of the study design (2 arms: d-cycloserine 250mg vs. placebo - twice daily for 4 weeks). Since the study went on to change design and then terminate prior to completing accrual, it is not useful to report baseline measures by the original arms/groups.
Arm/Group | All Participants (Original Version)
Number analyzed (Participants) | 7
Age, Customized [Number; unit: participants]
  40-50 years | 1
  51-60 years | 2
  61-70 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Difference in Patient-reported Pain Intensity Scores Between the 3 Arms After the Treatment Period Using the Brief Pain Inventory
Description: Compare patient-reported pain intensity scores after the treatment period (12 weeks) between the 3 arms of the trial.
Time Frame: From the date that the first patient is registered until the last patient completes the 12 weeks of study intervention (approximately 1 year)
Population: No patients were analyzed for this outcome measure due to a change in study design followed by early termination of the study.
Groups:
- Placebo (Revised Version): Placebo administered orally at a dose of twice per day for 4 weeks.
Arm/Group | D-cycloserine 250mg | Placebo (Original Version) | D-cycloserine 200mg | D-cycloserine 50 mg | Placebo (Revised Version)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Change in Individual Patients' Self-reported Overall Pain Relief Scores Before and After the Treatment Period
Description: Compare individual patients' self-reported pain relief scores before and after the treatment period.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | D-cycloserine 250mg | Placebo (Original Version) | D-cycloserine 200mg | D-cycloserine 50 mg | Placebo (Revised Version)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in Neuropathic Pain Scores in and Between Study Arms Using the Neuropathic Pain Inventory, the FACT-Taxane, and the Leonard Scale.
Description: Compare changes in neuropathic pain scores within each arm, as well as between the 3 arms of the study. Neuropathic pain will be assessed using 3 tools: the Neuropathic Pain Inventory, the FACT-Taxane, and the Leonard Scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | D-cycloserine 250mg | Placebo (Original Version) | D-cycloserine 200mg | D-cycloserine 50 mg | Placebo (Revised Version)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Differences in Pain Interference Between Study Arms Using the Brief Pain Inventory and the FACT-Taxane
Description: Compare the pain interference scores after study treatment between study arms using the brief pain inventory and the FACT-Taxane.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | D-cycloserine 250mg | Placebo (Original Version) | D-cycloserine 200mg | D-cycloserine 50 mg | Placebo (Revised Version)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Change in the Amount of Opioid Medication Used by Patients in Each Arm Before and After Study Treatment
Description: Record the amount of opioid medication used by patients in each arm before and after the study treatment period.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | D-cycloserine 250mg | Placebo (Original Version) | D-cycloserine 200mg | D-cycloserine 50 mg | Placebo (Revised Version)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo (Original Version) | D-cycloserine 250mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Early termination resulted from a change in funding source (which ultimately fell through) along with drug manufacturing delays. Data could not be analyzed based on only 7 patients, all of whom were enrolled under the original design version.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes